CLINICAL TRIAL: NCT00397917
Title: Oral Cleft Prevention Program
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Iowa (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); RTI International (Other); University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Jeff Murray, Professor of Pediatrics, University of Iowa
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NIDCR-17958; U01DE017958 (NIH)
Record Dates: First submitted 2006-11-08; First posted 2006-11-10 (Estimated); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Cleft Lip; Cleft Palate
MeSH Terms: conditions — Cleft Lip; Cleft Palate | interventions — Folic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Random number assignments
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 400 micrograms of folic acid (Active Comparator): Blinded study with two arms one of 400ug in arm 1
  Interventions: Drug: Folic acid: 4 mg versus 0.4 mg per day
- 4mg of folic acid (Active Comparator): Second arm is 4mg of folic acid in arm 2
  Interventions: Drug: Folic acid: 4 mg versus 0.4 mg per day

INTERVENTIONS:
Drug: Folic acid: 4 mg versus 0.4 mg per day — Folic acid

SUMMARY:
The purpose of this study is to asses if taking 4 mg of folic acid per day at preconception and during the first three months of pregnancy decreases the risk of having a child with cleft lip and palate compared to 0.4 mg folic acid for women who have an oral cleft or have had previously child with an oral cleft.

DETAILED DESCRIPTION:
Cleft lip and palate is a common and burdensome birth defect that has large health ramifications and requires surgical, speech, behavioral, dental, and medical interventions. There is some evidence suggesting that taking folic acid particularly at large doses during preconception and first trimester of pregnancy may decrease the risk of oral cleft recurrence, which is the risk of having a child with an oral cleft for women who have an oral cleft or who have had a child with a cleft. However this evidence is based on study designs that are incapable of contributing the preventive effects to folic acid with adequate confidence, and the real effect of folic acid on cleft recurrence prevention remains to be identified. Taking 4 mg of folic acid per day at preconception and first trimester of pregnancy has also been shown to prevent the recurrence of neural tube defects by up to 70%, providing further support to evaluate this intervention for oral cleft recurrence.

This study evaluates the effects of supplementation with 4 versus 0.4 mg of folic acid per day at preconception and during the first three months of pregnancy on recurrence of cleft lip and palate. Up to 6000 women will be randomly assigned to 4 versus 0.4 mg groups. The primary aim is to compare the recurrence rates in the offspring of trial mothers in the two groups. Secondary aims are to compare the two groups on several outcomes including miscarriage, twinning, pre-eclampsia, serum and red cell folate levels, severity of oral clefts and occurrence of other birth defects in the offspring of trial mothers, and birth weight and gestational age of trial babies, and to compare the recurrence in the two groups to that in historic controls.

ELIGIBILITY:
Inclusion Criteria:

* Women with cleft lip with/out palate (CLP), 16 to 45 years of age registered at the study clinics in Brazil or Women (16 to 45 years of age) with at least one natural child of any age with CLP registered at the study clinics.
* Women must reside in the catchment area of the study, which includes the states where the study clinics are located and surrounding states.

Exclusion Criteria:

* Consanguineous couples (up to third degree, i.e. first cousins or closer).
* Pregnany at the time of recruitment. Women will be recontacted later at an appropriate time for participation in the study.
* Couples either one of which have been sterilized.
* Taking any form of seizure medication.
* Planning to move outside of the study catchment area within the next year.
* B12 deficiency (<174 pg/mL or 129.15 pmol/L).
* Being allergic to folic acid.

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4000 (Actual)
Dates: Start 2006-11; Primary Completion 2012-05 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Recurrence of cleft lip and palate | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Murray, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No
Individual level data will not be shared unless de-identified

REFERENCES:
- [Result] Vila-Nova C, Wehby GL, Queiros FC, Chakraborty H, Felix TM, Goco N, Moore J, Gewehr EV, Lins L, Affonso CM, Murray JC. Periconceptional use of folic acid and risk of miscarriage - findings of the Oral Cleft Prevention Program in Brazil. J Perinat Med. 2013 Jul;41(4):461-6. doi: 10.1515/jpm-2012-0173. PMID 23669628
- [Derived] Wehby GL, Goco N, Moretti-Ferreira D, Felix T, Richieri-Costa A, Padovani C, Queiros F, Guimaraes CV, Pereira R, Litavecz S, Hartwell T, Chakraborty H, Javois L, Murray JC. Oral cleft prevention program (OCPP). BMC Pediatr. 2012 Nov 26;12:184. doi: 10.1186/1471-2431-12-184. PMID 23181832